CLINICAL TRIAL: NCT05041946
Title: Patient Controlled Methylphenidate for Cancer Related Fatigue: A Double Blind, Randomized, Placebo Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-0537; NCI-2021-10777 (Other: NCI ID)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Fatigue; Cancer
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Methylphenidate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate (Experimental): treatment of attention deficit disorder and narcolepsy (sleep disorder)
  Interventions: Drug: Methylphenidate; Other: Placebo (Sugar Pill)
- Placebo (Experimental): Sugar pill
  Interventions: Drug: Methylphenidate; Other: Placebo (Sugar Pill)

INTERVENTIONS:
Drug: Methylphenidate — Given PO
Other: Placebo (Sugar Pill) — Given PO

SUMMARY:
To determine the effectiveness of patient controlled methylphenidate as compared to placebo for the management of cancer related fatigue as determined by the Functional Assessment of Chronic Illness Therapy (FACIT)-F Fatigue score.

DETAILED DESCRIPTION:
Primary objective:

-To determine the effectiveness of patient controlled methylphenidate as compared to placebo for the management of cancer related fatigue as determined by the Functional Assessment of Chronic Illness Therapy (FACIT)-F Fatigue score

Secondary objective

* To assess the efficacy of as needed methylphenidate on pain, sedation and quality of life.
* To assess the potential side effects of methylphenidate on appetite, insomnia and anxiety

ELIGIBILITY:
Inclusion Criteria:

* Presence of fatigue on a numerical scale during the last 24 hours of more or equal to 4 on a 0 to 10 scale in which 0 equals no fatigue and 10 worst possible fatigue.
* Patients should describe fatigue as being present for a minimum of four days.
* If patients are on opioids for the treatment of cancer pain, change of opioids is allowed.
* No clinical evidence of cognitive failure, with normal Mini Mental State Examination (MMSE). A score of 24 is considered as normal.
* Sign written informed consent.
* Patients must be 18 years or older.
* Patient willing to keep a daily diary, engage in daily telephone follow up with a nurse, and after 7 days of treatment patient will return for a follow up visit.
* Patient must have telephone access to be contacted daily by the research nurse.
* Hemoglobin of >/=10 g/dl within 2 weeks of enrollment. If the patient has not had blood drawn for a hemoglobin level in the past two weeks, one will be done to determine the eligibility.

Exclusion Criteria:

* Major contraindication to methylphenidate i.e. hypersensitivity, anxiety, tension, agitation, or motor tics
* Currently on methylphenidate or has been on methylphenidate within the last 10 days.
* Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study.
* Pregnant or lactating women.
* Patients taking MAO inhibitors, tricyclic antidepressants and clonidine.
* Patients with glaucoma, history of marked anxiety disorder, or history of substance abuse.
* CAGE questionnaire score for the last 2 years is 2 or above on a 0 to 4 scale
* History of Tourette's syndrome
* Patients with tachycardia and uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-07-16 (Actual); Primary Completion 2004-12-15 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
To establish the effectiveness of patient the management of cancer related fatigue as determined by the Functional Assessment of Chronic Illness Therapy (FACIT)-F Fatigue score: 0-10 numerical scale. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org